CLINICAL TRIAL: NCT00617903
Title: A 12-week Exploratory, Multicenter, Double-blind, Vehicle-controlled Study to Investigate the Efficacy and Safety of Topical Azelaic Acid 15% Foam Twice Daily in Patients With Papulopustular Rosacea
Brief Title: Exploration of Safety and Efficacy of AzA 15% Foam Twice a Day in Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1402140
Record Dates: First submitted 2008-01-22; First posted 2008-02-18 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2013-12

CONDITIONS: Papulopustular Rosacea
Keywords: rosacea; papulopustular; azelaic acid; foam
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic acid foam, 15% (BAY39-6251) (Experimental): Participants received azelaic acid foam, 15% topically twice daily for 12 weeks
  Interventions: Drug: Azelaic acid
- Vehicle foam (Placebo Comparator): Participants received vehicle foam topically twice daily for 12 weeks
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Azelaic acid — 15% foam to be applied topically twice daily
  Arms: Azelaic acid foam, 15% (BAY39-6251)
Drug: Vehicle foam — Active-ingredient-free vehicle to be applied topically twice daily
  Arms: Vehicle foam

SUMMARY:
This exploratory study is being performed to determine whether a new form formulation of azelaic acid 15% is effective in the treatment of papulopustular rosecea.

ELIGIBILITY:
Inclusion Criteria:

* male and female patient at least 18 years of age
* signed informed consent
* Papulopustular rosacea with a minimum of 10 and a maximum of 50 papules and/or pustules, persistent erythema, and telangiectasia
* Ability and willingness to accept and comply with treatment and required medical examinations

Exclusion Criteria:

* Known non-responders to azelaic acid
* Erythematotelangiectatic, rhinophymatous, ocular, or steroid rosacea
* Presence of dermatoses that could interfere with the rosacea diagnosis
* Treatment with isotretinoin in the six months prior to randomization
* Treatment of the face with topical retinoids during the two weeks prior to randomization
* Treatment with oral antibiotics during the four weeks prior to randomization
* Treatment with topical antibiotics
* Treatment with systemic corticosteroids during 4 weeks prior to randomization
* Treatment of the face with topical corticosteroids during 2 weeks prior to randomization
* Treatment of the face with topical imidazole antimycotics during 2 weeks prior to randomization
* Treatment of the face with topical azelaic acid formulations during 2 weeks prior to randomization
* Use of a sauna during 2 weeks prior to randomization and during the study
* Facial laser surgery for telangiectasia during 6 weeks prior to randomization
* Planned concurrent use of any treatment other than study medication that affects rosacea
* History of hypersensitivity to propylene glycol or any other ingredient of the study drugs
* Participation in another clinical trial during the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (7):
  - Denver, Colorado
  - Olathe, Kansas
  - Henderson, Nevada
  - Albuquerque, New Mexico
  - Mason, Ohio
  - Austin, Texas
  - Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Started | 41 | 42
Completed | 38 | 35
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.9) | 51.5 (12.5) | 50.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 16 | 19 | 35
Previous duration of rosacea [Mean (Standard Deviation); unit: Months] | 88.5 (63.8) | 91.9 (77.0) | 90.2 (70.4)
Investigator's Global Assessment (IGA) score at Baseline [Mean (Standard Deviation); unit: Scores on a scale] — IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3- Mild to Moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe / Therapeutic success is defined as an IGA score of clear or minimal (0 to 1).
  Scores on a scale | 4.0 (0.9) | 3.9 (0.9) | 3.9 (0.9)
Number of inflammatory lesions per participant at Baseline [Mean (Standard Deviation); unit: Inflammatory lesions] | 18.0 (10.61) | 17.6 (8.36) | 17.8 (9.48)
Erythema intensity score at baseline [Mean (Standard Deviation); unit: Scores on a scale] — Erythema intensity score: 1 - Clear or almost clear; 2 - Mild; 3 - Moderate; 4 - Severe
  Scores on a scale | 3.1 (0.5) | 3.0 (0.5) | 3.0 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Nominal Change From Baseline in Inflammatory Lesion (IL) Count (Sum of Papules and Pustules) Per Participant at End of Study (LOCF: Last Observation Carried Forward)
Time Frame: Baseline and End of Study (Week 12)
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Inflammatory lesions | -11.7 (8.53) | -10.8 (7.80)

2. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Therapeutic Success at End of Study (LOCF)
Description: IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3- Mild to Moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe / Therapeutic success is defined as an IGA score of clear or minimal (0 to 1).
Time Frame: At End of Study (Week 12)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants | 46.3 | 47.6

3. Primary Outcome: Grouped Change From Baseline in Erythema Intensity Score at End of Study (LOCF)
Description: Erythema intensity score: 1 - Clear or almost clear; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: Baseline and End of Study (Week 12)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Improved | 61.0 | 47.6
  No change | 36.6 | 45.2
  Worse | 2.4 | 7.1

4. Secondary Outcome: Mean of Inflammatory Lesion Count Per Participant at Weeks 4, 8, 12 and End of Study (LOCF)
Time Frame: At Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Inflammatory lesions
  Week 4 | 9.1 (7.93) | 11.7 (9.23)
  Week 8 | 6.8 (7.59) | 6.6 (5.57)
  Week 12 | 4.3 (5.86) | 4.6 (5.47)
  End of Study | 6.3 (10.64) | 6.8 (8.46)

5. Secondary Outcome: Nominal Change From Baseline in Inflammatory Lesion Count Per Participant at Weeks 4, 8 and 12
Time Frame: Baseline and Weeks 4, 8 and 12
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Inflammatory lesions
  Week 4 | -7.5 (4.68) | -5.8 (4.95)
  Week 8 | -9.9 (5.88) | -10.3 (6.62)
  Week 12 | -12.4 (8.38) | -12.4 (7.26)

6. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count Per Participant at Weeks 4, 8, 12 and End of Study (LOCF)
Time Frame: Baseline and Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Mean (Standard Deviation); unit: Percent change in Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percent change in Inflammatory lesions
  Week 4 | -49.5 (23.68) | -37.7 (36.70)
  Week 8 | -62.7 (29.82) | -62.8 (27.71)
  Week 12 | -75.1 (33.80) | -74.8 (32.40)
  End of Study | -71.2 (36.42) | -65.3 (40.11)

7. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: as for outcome 2
Time Frame: At Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4-clear | 0 | 2.6
  Week 4-minimal | 20.5 | 10.5
  Week 4-mild | 17.9 | 21.1
  Week 4-mild to moderate | 23.1 | 21.1
  Week 4-moderate | 30.8 | 26.3
  Week 4-moderate to severe | 7.7 | 13.2
  Week 4-severe | 0 | 5.3
  Week 8-clear | 7.9 | 8.1
  Week 8-minimal | 28.9 | 27.0
  Week 8-mild | 18.4 | 16.2
  Week 8-mild to moderate | 21.1 | 16.2
  Week 8-moderate | 15.8 | 21.6
  Week 8-moderate to severe | 7.9 | 8.1
  Week 8-severe | 0 | 2.7
  Week 12-clear | 10.5 | 17.1
  Week 12-minimal | 36.8 | 37.1
  Week 12-mild | 26.3 | 8.6
  Week 12-mild to moderate | 21.1 | 20.0
  Week 12-moderate | 0 | 8.6
  Week 12-moderate to severe | 5.3 | 8.6
  Week 12-severe | 0 | 0
  End of Study-clear | 9.8 | 16.7
  End of Study-minimal | 36.6 | 31.0
  End of Study-mild | 24.4 | 7.1
  End of Study-mild to moderate | 19.5 | 19.0
  End of Study-moderate | 0 | 11.9
  End of Study-moderate to severe | 7.3 | 14.3
  End of Study-severe | 2.4 | 0

8. Secondary Outcome: Change From Baseline in IGA Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: as for outcome 2
Time Frame: Baseline and Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Scores on a scale
  Week 4 | -1.0 (1.2) | -0.7 (1.1)
  Week 8 | -1.6 (1.3) | -1.3 (1.4)
  Week 12 | -2.1 (1.2) | -1.9 (1.3)
  End of Study | -2.0 (1.3) | -1.7 (1.4)

9. Secondary Outcome: Percentage of Participants With Erythema Intensity Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: Erythema intensity score: 1 - Clear or almost clear; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: At Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4-clear or almost clear | 5.1 | 0
  Week 4-mild | 30.8 | 42.1
  Week 4-moderate | 51.3 | 50.0
  Week 4-severe | 12.8 | 7.9
  Week 8-clear or almost clear | 13.2 | 10.8
  Week 8-mild | 36.8 | 32.4
  Week 8-moderate | 42.1 | 45.9
  Week 8-severe | 7.9 | 10.8
  Week 12-clear or almost clear | 18.4 | 25.7
  Week 12-mild | 42.1 | 22.9
  Week 12-moderate | 34.2 | 45.7
  Week 12-severe | 5.3 | 5.7
  End of Study-clear or almost clear | 17.1 | 21.4
  End of Study-mild | 41.5 | 21.4
  End of Study-moderate | 34.1 | 52.4
  End of Study-severe | 7.3 | 4.8

10. Secondary Outcome: Change From Baseline in Erythema Intensity Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: Erythema intensity score: 1 - Clear or almost clear; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: Baseline and Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Scores on a scale
  Week 4 | -0.3 (0.6) | -0.4 (0.6)
  Week 8 | -0.6 (0.7) | -0.5 (0.8)
  Week 12 | -0.8 (0.8) | -0.7 (1.0)
  End of Study | -0.8 (0.8) | -0.6 (0.9)

11. Secondary Outcome: Grouped Change From Baseline in Erythema Intensity Score at Weeks 4, 8 and 12
Description: Erythema intensity score: 1 - Clear or almost clear; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: Baseline and Weeks 4, 8 and 12
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4-Improved | 35.9 | 42.1
  Week 4-No change | 59.0 | 52.6
  Week 4-Worse | 5.1 | 5.3
  Week 8-Improved | 50.0 | 48.6
  Week 8-No change | 50.0 | 40.5
  Week 8-Worse | 0 | 10.8
  Week 12-Improved | 63.2 | 54.3
  Week 12-No change | 34.2 | 37.1
  Week 12-Worse | 2.6 | 8.6

12. Secondary Outcome: Percentage of Participants With Telangiectasia Intensity Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: Telangiectasia intensity score: 1 - None; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: At Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4-none | 0 | 2.6
  Week 4-mild | 35.9 | 42.1
  Week 4-moderate | 64.1 | 55.3
  Week 4-severe | 0 | 0
  Week 8-none | 0 | 5.4
  Week 8-mild | 42.1 | 56.8
  Week 8-moderate | 57.9 | 37.8
  Week 8-severe | 0 | 0
  Week 12-none | 2.6 | 2.9
  Week 12-mild | 42.1 | 62.9
  Week 12-moderate | 55.3 | 34.3
  Week 12-severe | 0 | 0
  End of Study-none | 2.4 | 2.4
  End of Study-mild | 41.5 | 59.5
  End of Study-moderate | 56.1 | 38.1
  End of Study-severe | 0 | 0

13. Secondary Outcome: Change From Baseline in Telangiectasia Intensity Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: Telangiectasia intensity score: 1 - None; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: Baseline and Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Scores on a scale
  Week 4 | 0.0 (0.3) | -0.1 (0.4)
  Week 8 | -0.1 (0.3) | -0.3 (0.5)
  Week 12 | -0.2 (0.4) | -0.3 (0.5)
  End of Study | -0.1 (0.4) | -0.2 (0.4)

14. Secondary Outcome: Grouped Change From Baseline in Telangiectasia Intensity Scores at Weeks 4, 8, 12 and End of Study (LOCF)
Description: Telangiectasia intensity score: 1 - None; 2 - Mild; 3 - Moderate; 4 - Severe
Time Frame: Baseline and Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4-Improved | 5.1 | 10.5
  Week 4-No change | 92.3 | 86.8
  Week 4-Worse | 2.6 | 2.6
  Week 8-Improved | 10.5 | 27.0
  Week 8-No change | 89.5 | 73.0
  Week 8-Worse | 0 | 0
  Week 12-Improved | 15.8 | 28.6
  Week 12-No change | 84.2 | 71.4
  Week 12-Worse | 0 | 0
  End of Study-Improved | 14.6 | 23.8
  End of Study-No change | 85.4 | 76.2
  End of Study-Worse | 0 | 0

15. Secondary Outcome: Investigator's Rating of Overall Improvement at End of Study
Description: Investigator's rating of overall improvement: 1 - excellent improvement; 2 - marked improvement; 3 - moderate improvement; 4 - no change; 5 - deterioration
Time Frame: At End of Study (Week 12)
Population: All subjects of the FAS population for which this measurement was evaluated (one-time evaluation at the last study visit; FAS observed cases)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 38 | 40
Percentage of participants
  Excellent Improvement | 34.2 | 40.0
  Marked Improvement | 23.7 | 17.5
  Moderate Improvement | 31.6 | 27.5
  No Improvement | 7.9 | 12.5
  Deterioration | 2.6 | 2.5

16. Secondary Outcome: Patients' Rating of Overall Improvement at End of Study
Description: Patient's rating of overall improvement: 1 - excellent; 2 - good; 3 - fair; 4 - no improvement; 5 - worse
Time Frame: At End of Study (Week 12)
Population: All subjects of the FAS population for which this measurement was evaluated (one-time evaluation at the last study visit; FAS observed cases
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 38 | 40
Percentage of participants
  Excellent Improvement | 36.8 | 27.5
  Good Improvement | 28.9 | 22.5
  Fair Improvement | 21.1 | 22.5
  No Improvement | 5.3 | 20.0
  Worse | 7.9 | 7.5

17. Secondary Outcome: Patients' Opinion on Cosmetic Acceptability at End of Study
Description: Patient's opinion on cosmetic acceptability: 1 - very good; 2 - good; 3 - satisfactory; 4 - poor; 5 - no opinion
Time Frame: At End of Study (Week 12)
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 38 | 40
Percentage of participants
  Very Good | 42.1 | 35.0
  Good | 36.8 | 37.5
  Satisfactory | 10.5 | 5.0
  Poor | 5.3 | 10.0
  No Opinion | 5.3 | 12.5

18. Secondary Outcome: Percentage of Participants With IGA Based Therapeutic Success at Weeks 4, 8 and 12
Description: IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3- Mild to Moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe / Therapeutic success was defined as an IGA score of clear or minimal (0 to 1).").
Time Frame: At Weeks 4, 8 and 12
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4 | 20.5 | 13.2
  Week 8 | 36.8 | 35.1
  Week 12 | 47.4 | 54.3

19. Secondary Outcome: Percentage of Participants With IGA Based Patient Response at Weeks 4, 8, 12 and End of Study (LOCF)
Description: IGA based Patient response was defined as an IGA score of clear, minimal or mild (0, 1, 2).
Time Frame: At Weeks 4, 8, 12 and End of Study (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 41 | 42
Percentage of participants
  Week 4 | 38.5 | 34.2
  Week 8 | 55.3 | 51.4
  Week 12 | 73.7 | 62.9
  End of Study | 70.7 | 54.8

ADVERSE EVENTS:
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 14/41 | 10/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Foam, 15% (BAY39-6251) (N=41) | Vehicle Foam (N=42)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Administration site reaction (General disorders) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 4 (4) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A) Investigator shall provide Sponsor with intended publication 60 days upfront publication date, Sponsor has 30 d to comment, recommended changes shall not be unreasonably refused B) Sponsor has the right to ask Investigator to delay publication for a maximum of 90 days C) Investigative data will be pooled and published by Sponsor - no other publication without the consent of all parties prior to publication of the pooled data, or within 12 months after LPLV, whatever comes first